CLINICAL TRIAL: NCT02981108
Title: A Phase 1/2, Open-label, Multicenter Study to Evaluate Safety, Tolerability, Pharmacokinetics and Efficacy of HS-10296 in Patients With Locally Advanced or Metastatic Non-Small-Cell Lung Cancer
Brief Title: A Study to Evaluate Safety, PK and Efficacy of HS-10296 in Patients With NSCLC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10296-12-01
Record Dates: First submitted 2016-11-28; First posted 2016-12-02 (Estimated); Results first posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2022-12

CONDITIONS: Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Escalation Cohort 1 (Experimental): Oral Once-Daily Administration of HS-10296 55mg
  Interventions: Drug: HS-10296
- Escalation Cohort 2 (Experimental): Oral Once-Daily Administration of HS-10296 110mg
  Interventions: Drug: HS-10296
- Escalation Cohort 3 (Experimental): Oral Once-Daily Administration of HS-10296 220mg
  Interventions: Drug: HS-10296
- Escalation Cohort 4 (Experimental): Oral Once-Daily Administration of HS-10296 260mg
  Interventions: Drug: HS-10296
- Expansion Cohort 1 (Experimental): Oral Once-Daily Administration of HS-10296 55mg
  Interventions: Drug: HS-10296
- Expansion Cohort 2 (Experimental): Oral Once-Daily Administration of HS-10296 110mg
  Interventions: Drug: HS-10296
- Expansion Cohort 3 (Experimental): Oral Once-Daily Administration of HS-10296 220mg
  Interventions: Drug: HS-10296
- Phase 2 Extension (Experimental): Oral Once-Daily Administration of HS-10296 110mg (RP2D)
  Interventions: Drug: HS-10296

INTERVENTIONS:
Drug: HS-10296 — HS-10296: 5-, 10-, 40-, and 55-mg tablet, immediate-release formulation. Patients should avoid consumption of food for at least 1 hour prior to and 2 hours post dosing. RP2D is determined at 110 mg QD.

SUMMARY:
This is a Phase 1/2, open-label, multicenter study of HS-10296 with dose escalation, dose expansion and extension cohorts in locally advanced or metastatic non-small-cell lung cancer (NSCLC) patients who have progressed following prior therapy with an epidermal growth factor receptor(EGFR) tyrosine kinase inhibitor (TKI) agent. The study is designed to evaluate safety, tolerability, pharmacokinetics (PK), and anti-tumor activity of once-daily and orally (PO) administered HS-10296. The overall study design is shown in the flow chart below, which consists of 3 phases: dose escalation, dose expansion and extension cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated written informed consent prior to any study-specific procedures, sampling, and analyses. If a patient declines to participate in any voluntary exploratory research and/or genetic component of the study, there will be no penalty or loss of benefit to the patient and he/she will not be excluded from other aspects of the study.
2. Age at least 18 years.
3. Histological or cytological confirmation diagnosis of NSCLC.
4. Radiological documentation of disease progression while on a previous continuous treatment with an EGFR TKI, e.g., gefitinib or erlotinib. In addition, other lines of therapy may have been given. All patients must have documented radiological progression on the last treatment administered, prior to enrolling in the study.
5. Patients must fulfill one of the following:

   * Confirmation that the tumor harbors an EGFR mutation known to be associated with EGFR TKI sensitivity (including G719X, exon 19 deletion, L858R, L861Q) OR must have experienced clinical benefit from EGFR TKI, according to the Jackman criteria (followed by systemic objective progression (RECIST or World Health Organization [WHO]) while on continuous treatment with an EGFR TKI.
6. For the dose expansion and extension cohorts, patients also must have confirmation of tumor T790M+ mutation status from a biopsy sample taken after disease progression on the most recent treatment regimen with an EGFR TKI.

   Prior to entry, a result from the central analysis of the patient's T790M mutation status must be obtained.
7. World Health Organization (WHO) performance status equal to 0-1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.
8. At least 1 lesion that has not previously been irradiated, that has not been chosen for biopsy during the study Screening period,and that can be accurately measured at Baseline as ≥ 10mm in the longest diameter (except lymph nodes which must have short axis ≥ 15mm) with computerized tomography (CT) or magnetic resonance imaging (MRI), which is suitable for accurately repeated measurements.
9. Females of child-bearing potential should be using adequate contraceptive measures throughout the study, should not be breast feeding at the time of screening, during the study and until 3 months after completion of study, and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling 1 of the following criteria at screening:

   * Post-menopausal defined as age more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
   * Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more, following cessation of exogenous hormonal treatments, and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range for the laboratory.
   * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not by tubal ligation.
10. Male patients should be willing to use barrier contraception (i.e., condoms).
11. For the dose expansion paired biopsy cohort:

    * Presence of at least 1 non-target lesion suitable for multiple biopsies while on treatment.
12. For inclusion in optional genetic research, the patient must provide a written informed consent for genetic research.

Exclusion Criteria:

1. Treatment with any of the following:

   * An EGFR TKI (e.g., erlotinib, gefitinib, or osimertinib) within 8 days or approximately 5 times the half-life of the specific drug, whichever is longer, of the first dose of study treatment. (If sufficient wash-out time has not occurred due to scheduling or PK properties, an alternative appropriate wash-out time based on known duration and time to reversibility of drug-related adverse events must be agreed upon by Hansoh and the Investigator).
   * Any cytotoxic chemotherapy, investigational agents, or anticancer drugs for advanced NSCLC used for a previous treatment regimen or clinical study within 14 days of the first dose of study treatment.
   * Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study treatment.
   * Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment, with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation which must be completed within 4 weeks of the first dose of study treatment.
2. Previously untreated NSCLC patients. To be eligible for this study, patients must have received and progressed on EGFR TKI therapy.
3. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE), Grade 1, at the time of starting study treatment with the exception of alopecia and Grade 2, prior platinum-therapy related neuropathy.
4. Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least 4 weeks prior to start of study treatment.
5. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension or active bleeding diatheses, which, in the Investigator's opinion, makes it undesirable for the patient to participate in the trial OR which would jeopardize compliance with the protocol such as active infection (e.g., hepatitis B, hepatitis C or human immunodeficiency virus [HIV]). Screening for chronic conditions is not required.
6. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 electrocardiograms (ECGs), using the Screening clinic ECG machine and Fridericia's formula for QT interval correction.
   * Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval >250msec).
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval.
7. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
8. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

   * Absolute neutrophil count < 1.5 x 109/L.
   * Platelet count < 100 x 109/L.
   * Hemoglobin < 90 g/L (< 9 g/dL).
   * Alanine aminotransferase > 2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or > 5 times the ULN in the presence of liver metastases.
   * Aspartate aminotransferase > 2.5 times the ULN if no demonstrable liver metastases or > 5 times the ULN in the presence of liver metastases.
   * Total bilirubin > 1.5 times the ULN if no liver metastases or > 3 times the ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases.
   * Creatinine > 1.5 times the ULN concurrent with creatinine clearance < 50 mL/min (measured or calculated by the Cockcroft - Gault equation); confirmation of creatinine clearance is only required when creatinine is > 1.5 times the ULN.
9. Refractory nausea, vomiting, or chronic gastrointestinal diseases, inability to swallow the study medication, or previous significant bowel resection that would preclude adequate absorption of HS-10296.
10. History of hypersensitivity to any active or inactive ingredient of HS-10296 or to a drug with a similar chemical structure or class to HS-10296.
11. Women who are breast feeding.
12. Involvement in study planning and conduct (i.e., Hansoh staff or staff at the study site).
13. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
14. Any disease or condition that, in the opinion of the Investigator, would compromise the safety of the patient or interfere with study assessments.
15. The following are considered criteria for exclusion from the exploratory genetic research:

    * Previous allogenic bone marrow transplant.
    * Non-leukocyte leukocyte-depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2019-01-05 (Actual); Study Completion 2023-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Beverly Hills Cancer Center, Beverly Hills, California
  - University of California San Diego Medical Center Moores Cancer Center, San Diego, California
  - University of Colorado-1775 Aurora Court, Aurora, Colorado
  - Sylvester Comprehensive Cancer Center, Deerfield Beach, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Baptist Healthcare Systems Inc. Baptist Health Floyd, New Albany, Indiana
  - Dartmouth-Hitchcock Medical Center, Hanover, New Hampshire
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - MultiCare Institute for Research and Innovation, Tacoma, Washington

REFERENCES:
- [Derived] Yang JC, Camidge DR, Yang CT, Zhou J, Guo R, Chiu CH, Chang GC, Shiah HS, Chen Y, Wang CC, Berz D, Su WC, Yang N, Wang Z, Fang J, Chen J, Nikolinakos P, Lu Y, Pan H, Maniam A, Bazhenova L, Shirai K, Jahanzeb M, Willis M, Masood N, Chowhan N, Hsia TC, Jian H, Lu S. Safety, Efficacy, and Pharmacokinetics of Almonertinib (HS-10296) in Pretreated Patients With EGFR-Mutated Advanced NSCLC: A Multicenter, Open-label, Phase 1 Trial. J Thorac Oncol. 2020 Dec;15(12):1907-1918. doi: 10.1016/j.jtho.2020.09.001. Epub 2020 Sep 9. PMID 32916310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 364 patients were enrolled at 47 centers in 2 countries.
Groups:
- Phase 2 Extension: Oral Once-Daily Administration of HS-10296 (MTD or RP2D)
  HS-10296: HS-10296: 5-, 10-, 40-, and 55-mg tablet, immediate-release formulation. Patients should avoid consumption of food for at least 1 hour prior to and 2 hours post dosing. RP2D is determined at 110 mg QD.
Period: Overall Study
Arm/Group | Escalation Cohort 1 | Escalation Cohort 2 | Escalation Cohort 3 | Escalation Cohort 4 | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3 | Phase 2 Extension
Started | 6 | 6 | 8 | 6 | 30 | 33 | 31 | 244
Completed (Discontinuation of treatment) | 5 | 6 | 7 | 6 | 21 | 15 | 13 | 62
Not Completed | 1 | 0 | 1 | 0 | 9 | 18 | 18 | 182

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escalation Cohort 1 | Escalation Cohort 2 | Escalation Cohort 3 | Escalation Cohort 4 | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3 | Phase 2 Extension | Total
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 30 | 33 | 31 | 244 | 364
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 5 | 4 | 22 | 16 | 21 | 153 | 228
  >=65 years | 3 | 2 | 3 | 2 | 8 | 17 | 10 | 91 | 136
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 5 | 5 | 19 | 20 | 20 | 142 | 219
  Male | 1 | 3 | 3 | 1 | 11 | 13 | 11 | 102 | 145
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 6 | 7 | 5 | 29 | 31 | 31 | 244 | 358
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 4
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 7
  Taiwan | 5 | 6 | 5 | 5 | 13 | 17 | 18 | 55 | 124
  China | 0 | 0 | 1 | 0 | 16 | 14 | 13 | 189 | 233

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT) Phase I Part
Description: DLT is defined as one of the following HS-10296 related adverse event (AE) ：(1) Hematological toxicity ≥ Grade 4 neutropenia lasting more than 5 days, febrile neutropenia of any duration (absolute neutrophil count [ANC]) < 1.0 × 109/L and fever ≥ 38.5°C), Grade 4 thrombocytopenia, Grade 3 thrombocytopenia with bleeding, any requirement for platelet transfusion, Grade 4 anemia (unexplained by underlying disease); (2)Non-hematological toxicity ≥ CTCAE Grade 3 including Infection (including febrile neutropenia), confirmed prolongation of QT interval corrected with Fridericia's (QTcF) (> 500 ms absolute or > 60 ms above Baseline) and cardiac toxicity greater than Grade 3；(3)Any other toxicity that is greater than that at Baseline (clinically significant and/or unacceptable, and judged to be a DLT by the SRC), meets a protocol-defined stopping criteria (i.e., confirmed corneal ulceration), or results in a disruption of dosing schedule of more than 7 days.
Time Frame: 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Cohort 1 | Escalation Cohort 2 | Escalation Cohort 3 | Escalation Cohort 4
Number analyzed (Participants) | 6 | 6 | 8 | 6
Participants | 0 | 0 | 1 | 1

2. Primary Outcome: Overall Response Rate (ORR) Phase II Part
Description: ORR is defined as the percentage of patients with a complete response (CR) or partial response (PR) that was confirmed at a subsequent scan at least 6 weeks later, as assessed according to RECIST (Response Evaluation Criteria In Solid Tumors Criteria) version 1.1 for target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From the date of first dose until the date of disease progression or withdrawal from study, approximately 15 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 Extension
Number analyzed (Participants) | 244
percentage of participants | 65.6 [59.2 to 71.5]

3. Primary Outcome: Incidence and Severity of Adverse Events (AEs) Phase I Part
Description: An AE is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. An undesirable medical condition can be symptoms (e.g., nausea, chest pain), signs (e.g., tachycardia, enlarged liver), or the abnormal results of an investigation (e.g., laboratory findings, ECG). Any deterioration of the disease under study and associated symptoms or findings should not be regarded as an AE as far as the deterioration can be anticipated. The AE was graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0.
Time Frame: From the screening period to 28 days after treatment completion, approximately 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Cohort 1 | Escalation Cohort 2 | Escalation Cohort 3 | Escalation Cohort 4 | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 30 | 33 | 31
Participants
  At least one adverse event | 6 | 6 | 8 | 6 | 30 | 32 | 31
  At least one adverse event of Grade 3 or greater | 1 | 1 | 3 | 3 | 6 | 8 | 11
  At least one serious adverse event | 2 | 1 | 2 | 3 | 5 | 6 | 3

4. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of HS-10296 and HAS-719 From Zero to the 24-Hour Sampling Time (AUC0-24) After Single Dose of HS-10296
Description: Area under the plasma concentration versus time curve from time zero to the 24-hour sampling time at which the concentration was at or above the lower limit of quantification (LLQ). AUC0-24 was to be calculated according to the mixed log-linear trapezoidal rule.
Time Frame: From pre-dose to 24 hours after single dose on Day 1 of Cycle 0
Population: Data was collected for only Part 1 dose escalation Arms
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Escalation Cohort 1 | Escalation Cohort 2 | Escalation Cohort 3 | Escalation Cohort 4
Number analyzed (Participants) | 6 | 6 | 8 | 6
h*ng/mL
  HS-10296 | 1740.1175 (917.7303) | 5250.2364 (3345.8348) | 8174.4312 (8126.7012) | 8038.9348 (1648.4566)
  HAS-719 | 298.4934 (131.6189) | 696.4536 (293.4756) | 1152.1150 (475.5067) | 1564.3829 (488.6330)

5. Secondary Outcome: Elimination Half-life(T1/2) of HS-10296 and HAS-719
Description: Elimination half-life is the time measured for the concentration to decrease by one half. Half-life calculated by natural log 2 divided by λz.
Time Frame: From pre-dose to 120 hours after single dose on Day 1 of Cycle 0
Population: Data was collected for only Part 1 dose escalation Arms
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Escalation Cohort 1 | Escalation Cohort 2 | Escalation Cohort 3 | Escalation Cohort 4
Number analyzed (Participants) | 6 | 6 | 8 | 6
hours
  HS-10296 | 31.29 (9.57) | 30.62 (9.34) | 35.19 (13.89) | 34.81 (9.76)
  HAS-719 | 49.75 (10.70) | 55.36 (19.95) | 63.75 (29.83) | 57.79 (13.95)

6. Secondary Outcome: Css Max of HS-10296 and HAS-719 After Multiple Dose
Description: Observed maximum plasma concentration (Css max) after multiple dose of HS-10296 and HAS-719
Time Frame: From pre-dose to 21 days after multiple dose on Day 1 of Cycle 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Escalation Cohort 1 | Escalation Cohort 2 | Escalation Cohort 3 | Escalation Cohort 4 | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3 | Phase 2 Extension
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 30 | 33 | 31 | 244
ng/mL
  HS-10296 | 164.5000 (70.6222) | 352.8333 (102.7062) | 762.0000 (231.8888) | 765.4000 (285.2802) | 197.9308 (78.6513) | 413.2751 (194.0200) | 552.0635 (257.9572) | 352.5111 (185.3279)
  HAS-719 | 55.3500 (18.1391) | 118.1333 (26.9018) | 276.1667 (42.9391) | 338.2000 (119.3302) | 62.9535 (21.4094) | 142.1545 (49.4867) | 221.9404 (83.6900) | 118.3758 (43.3468)

7. Secondary Outcome: AUCss of HS-10296 and HAS-719 After Multiple Dose of HS-10296
Description: Area Under the Plasma Concentration Versus Time Curve at steady state (AUCss) of HS-10296 and HAS-719 after multiple dose of HS-10296
Time Frame: From pre-dose to 21 days after multiple dose on Day 1 of Cycle 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Escalation Cohort 1 | Escalation Cohort 2 | Escalation Cohort 3 | Escalation Cohort 4 | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3 | Phase 2 Extension
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 30 | 33 | 31 | 244
h*ng/mL
  HS-10296 | 2488.0953 (439.3443) | 7000.2498 (2832.8180) | 11994.8801 (3839.4164) | 14101.8608 (5294.1409) | 3550.8674 (1451.0173) | 7098.0738 (2826.1228) | 10185.6761 (4862.0070) | 6602.2491 (3482.0499)
  HAS-719 | 983.7103 (201.9267) | 2691.7220 (677.2407) | 5458.2304 (659.3078) | 8154.0849 (1144.0617) | 1304.4143 (429.1216) | 2852.8083 (820.1842) | 4692.6023 (1771.6881) | 2467.8527 (892.5071)

8. Secondary Outcome: Overall Response Rate (Phase I Part)
Description: as for outcome 2
Time Frame: From the date of first dose until the date of disease progression or withdrawal from study, approximately 15 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Escalation Cohort 1 | Escalation Cohort 2 | Escalation Cohort 3 | Escalation Cohort 4 | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 30 | 33 | 31
percentage of participants | 50.0 [11.8 to 88.2] | 66.7 [22.3 to 95.7] | 37.5 [8.5 to 75.5] | 16.7 [0.4 to 64.1] | 60.0 [40.6 to 77.3] | 54.5 [36.4 to 71.9] | 41.9 [24.5 to 60.9]

9. Secondary Outcome: Progression-free Survival (PFS)
Description: The PFS is defined as the time from date of first dosing until the date of objective disease progression as defined by Response Evaluation Criteria in Solid Tumors （RECIST） v1.1 or death (by any cause in the absence of progression) regardless of whether the patients withdraws from HS-10296 therapy or receives another anti-cancer therapy prior to progression. Progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From the date of enrollment until the date of disease progression or death from any cause, approximately 15 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Escalation Cohort 1 | Escalation Cohort 2 | Escalation Cohort 3 | Escalation Cohort 4 | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3 | Phase 2 Extension
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 30 | 33 | 31 | 244
months | 11.2 [3.0 to NA] — Since the curve that represents the upper confidence limits for the KM survivor function lies above 0.5, thus the upper limits for the median can not be estimated. | 7.0 [5.8 to 12.5] | 5.5 [1.1 to 8.4] | 3.7 [0.8 to 11.0] | 9.6 [6.7 to 15.1] | 13.6 [6.9 to 19.2] | 11.1 [8.3 to 24.8] | 12.4 [9.7 to 15.0]

10. Secondary Outcome: Disease Control Rate (DCR)
Description: Objective response is assessed by RECIST 1.1 thereby to evaluate disease control rate. The DCR is defined as the proportion of patients with a best overall response of CR, PR, or SD (stable disease).
Time Frame: From the date of first dose until the date of disease progression or withdrawal from study, approximately 15 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Escalation Cohort 1 | Escalation Cohort 2 | Escalation Cohort 3 | Escalation Cohort 4 | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3 | Phase 2 Extension
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 30 | 33 | 31 | 244
percentage of participants | 100.0 [54.1 to 100.0] | 100.0 [54.1 to 100.0] | 75.0 [34.9 to 96.8] | 50.0 [11.8 to 88.2] | 83.3 [65.3 to 94.4] | 97.0 [84.2 to 99.9] | 93.5 [78.6 to 99.2] | 93.4 [89.6 to 96.2]

11. Secondary Outcome: Overall Survival (OS) Phase II Part
Description: Overall survival will be assessed based on the date of first dose and survival status at the time of analysis. Overall survival is defined as the time from date of first dose until the documentation of death from any cause.
Time Frame: From the date of enrollment until the date of death from any cause, approximately 48 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Extension
Number analyzed (Participants) | 244
months | 31.5 [25.9 to 35.7]

12. Secondary Outcome: Depth of Response (DepOR)
Description: Depth of Response (DepOR) Only in part II dose-extention phase. DepOR is defined as the percentage change in tumor size, based on longest diameter or reconstructed volume, observed at the lowest point compared with baseline.
Time Frame: From the date of enrollment until the date of disease progression or death, approximately 15 months
Population: Based on the ICR evaluation results, DepOR analysis was performed on patients with efficacy evaluation
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Phase 2 Extension
Number analyzed (Participants) | 237
percentage of change from baseline | -47.89 (22.333)

13. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response (DoR) is defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression. The end of response should coincide with the date of progression or death from any cause used for the PFS endpoint. The time of the initial response will be defined as the latest of the dates contributing towards the first visit response of PR or CR. If a patient does not progress following a response, then DoR will be used as the PFS censoring time.
Time Frame: From the date of enrollment until the date of disease progression or death, approximately 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Escalation Cohort 1 | Escalation Cohort 2 | Escalation Cohort 3 | Escalation Cohort 4 | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3 | Phase 2 Extension
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 30 | 33 | 31 | 244
months | 13.9 [1.9 to NA] — Since the curve that represents the upper confidence limits for the KM survivor function lies above 0.5, thus the upper limits for the median can not be estimated. | 5.6 [4.2 to 9.5] | 5.6 [4.1 to 7.0] | 5.5 [NA to NA] — Since the curve that represents the upper confidence limits for the KM survivor function lies above 0.5, thus the upper limits for the median can not be estimated. | 8.3 [8.1 to 16.5] | 12.5 [5.5 to 22.1] | 22.1 [8.1 to 35.7] | 15.1 [12.9 to 16.6]

14. Secondary Outcome: Incidence and Severity of AEs Phase II Part
Description: as for outcome 3
Time Frame: From the screening period to 28 days after treatment completion, approximately 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Extension
Number analyzed (Participants) | 244
Participants
  At least 1 adverse event | 219
  At least one adverse event of Grade 3 or greater | 60
  At least one serious adverse event | 30

ADVERSE EVENTS:
Time Frame: Throughout the study, from informed consent until the end of the follow-up period. The follow-up period is defined as 28 ± 3 days after study treatment is discontinued, assessed up to 16 months. Deaths were assessed up to 48 months. Serious and Other (Non-Serious) Adverse Events were assessed up to 16 months.
Arm/Group | Escalation Cohort 1 | Escalation Cohort 2 | Escalation Cohort 3 | Escalation Cohort 4 | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3 | Phase 2 Extension
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/8 | 0/6 | 0/30 | 0/33 | 0/31 | 11/244
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/6 | 2/8 | 3/6 | 5/30 | 6/33 | 3/31 | 30/244
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 8/8 | 6/6 | 29/30 | 31/33 | 29/31 | 193/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Escalation Cohort 1 (N=6) | Escalation Cohort 2 (N=6) | Escalation Cohort 3 (N=8) | Escalation Cohort 4 (N=6) | Expansion Cohort 1 (N=30) | Expansion Cohort 2 (N=33) | Expansion Cohort 3 (N=31) | Phase 2 Extension (N=244)
Pneumonitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes ophthalmic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escalation Cohort 1 (N=6) | Escalation Cohort 2 (N=6) | Escalation Cohort 3 (N=8) | Escalation Cohort 4 (N=6) | Expansion Cohort 1 (N=30) | Expansion Cohort 2 (N=33) | Expansion Cohort 3 (N=31) | Phase 2 Extension (N=244)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 11 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 1 (1) | 7 (7)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (5)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 20 (20)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 5 (5) | 7 (7) | 11 (11)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 10 (10)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 4 (4) | 5 (5) | 15 (15)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 9 (9)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 3 (3) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 7 (7)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 3 (3) | 32 (32)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 2 (2) | 5 (5) | 28 (28)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Aspartate aminotransferase abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 2 (2) | 7 (7) | 33 (33)
Blood creatine phosphokinase MB increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 12 (12)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 11 (11)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myoglobin blood increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 3 (3) | 0 (0) | 14 (14)
Neutrophil percentage increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 3 (3) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 10 (10)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 7 (7) | 2 (2) | 2 (2) | 23 (23)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 11 (11)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 10 (10)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 10 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 8 (8) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Muscle spasticity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 17 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 6 (6) | 4 (4) | 7 (7) | 25 (25)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 6 (6) | 4 (4) | 28 (28)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 6 (6) | 6 (6) | 30 (30)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 6 (6)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT02981108/Prot_SAP_000.pdf